CLINICAL TRIAL: NCT00236288
Title: A Feasibility Study of Smoking Cessation Program in Radiation Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Walther Cancer Institute (Other)
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 0508-12; Walther Cancer Institute, Inc
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Cancer and Tobacco Abuse
Keywords: Cancer treatment and tobacco abuse
MeSH Terms: conditions — Neoplasms; Tobacco Use Disorder | interventions — Bupropion

INTERVENTIONS:
Drug: Bupropion and intensive behavioral therapy — To prescribe bupropion and behavioral therapy to patients and/or their families, who are currently receiving radiation.

SUMMARY:
To test the feasibility of an intensive behavioral and pharmacologic tobacco cessation program for radiation oncology patients and their families/companions.

DETAILED DESCRIPTION:
There is overwhelming evidence to support tobacco use as the number one cause of preventable cancer and cardiovascular death. Smoking is responsible for at least 30% of all cancer deaths and nearly 90% of lung cancer deaths. There is robust phase III randomized data to show improved smoking cessation with both behavioral strategies as well as pharmacologic interventions such as bupropion.

Despite significant evidence showing survival, toxicity and quality of life detriments in cancer patients who continue smoking after diagnosis, roughly one third of cancer patients continue to use tobacco. There is a relative paucity of data regarding smoking cessation programs in cancer patient populations. Several single institution, as well as cooperative group (ECOG), efforts have been published with varying results. However, to date, there are no published reports on the success of pharmacologic smoking cessation interventions in cancer patients.

Patients undergoing definitive/curative radiotherapy often receive daily treatment over the course of three to eight weeks. They are often accompanied and supported daily by family members or companions, many of whom smoke. This represents a huge exposure to the health care system and a unique opportunity for intensive intervention in both cancer patients and their families/companions during their "daily routine" of radiotherapy. To date, there is no published report on intensive tobacco cessation intervention concurrent with radiotherapy in cancer patients and their families or companions.

We propose a feasibility study of an intensive tobacco cessation program to be delivered to radiation oncology patients and/or their family/companions concurrent with planned radiotherapy. This program will feature an intensive behavioral intervention as well as the pharmacologic agent bupropion.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for Radiotherapy Patients
* age 18 years or older
* receiving three weeks or more of external beam radiotherapy
* report smoking one or more cigarettes in the past 30 days or self-identify as a smoker
* Cancer Stage:
* Stage I-III
* IVa Head and Neck Malignancy is allowed
* Stage I-IV breast, prostate, testis or lymphoma also allowed
* at least one year life expectancy
* have given written informed consent
* KPS 70-100

Eligibility for Family/Companions of Radiotherapy Patients (Note: Family members/companions are eligible for this protocol regardless of whether the index radiotherapy patient is eligible or willing to participate.)

* age 18 years or older
* at least one year life expectancy
* radiotherapy patient is receiving three weeks or more of external beam radiotherapy
* Person is committed to bringing/accompanying the patient to radiotherapy at least three days per week.
* report smoking one or more cigarettes in the past 30 days or self-identify as a smoker
* Family member/companion of patients under radiotherapy treatment for any stage of cancer
* have given written informed consent
* KPS 70-100

Exclusion Criteria:

* Exclusion Criteria for both Radiotherapy Patients and their Families/Companions
* serious or unstable cardiac, renal, hypertensive, pulmonary, endocrine, or neurologic disorders, as assessed by the study-site physician
* a current diagnosis of major depressive episode or a history of panic disorder, psychosis, bipolar disorder, or eating disorders
* pregnancy or lactation
* any history of allergy/intolerance or adverse reaction to bupropion
* history of seizure disorder, bulimia or anorexia nervosa
* use of an MAOi within 14 days
* current use of another antidepressant
* abrupt discontinuation of alcohol or sedatives
* unwilling/unable to meet with the behavioral interventionalist for 20 minutes, at least 3 days per week during the course of radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To test the feasibility of using the medication bupropion and behavioral therapy to help people stop smoking in the radiation oncology clinic. | 1 year from enrollment

SECONDARY OUTCOMES:
Smoking cessation status will be formally assessed by patient report, and for those reporting tobacco abstinence, confirmed by carbon monoxide breath testing concentrations of 10 ppm or less. | 1 year from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Anna McDaniel, DNS, RN, FAAN, Principal Investigator — Department of Environments for Health, Indiana University School of Nursing
Locations (1):
- Indiana University, Department of Radiation Oncology, Indianapolis, Indiana, United States